CLINICAL TRIAL: NCT04332757
Title: The Efficacy of a Post-Partum Physical Development Programme on Occupational Physical Performance and Musculoskeletal Health
Brief Title: Postpartum Exercise and Return to Fitness: Optimise Readiness for Military Mums (PERFORM)
Acronym: PERFORM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: University of Nottingham (Other); Robert Gordon University (Other); University of Stirling (Other); Ministry of Defence, United Kingdom (Other Government); Clare Pacey Physiotherapy Limited (Unknown)
Responsible Party: Principal Investigator, Craig Sale, Professor of Human Physiology, Director of the Sport, Health and Performance Enhancement Research Centre, Nottingham Trent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 349408; ASC/BA/00665 (Other Grant/Funding Number: ASC Contract Number)
Record Dates: First submitted 2020-03-24; First posted 2020-04-03 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Postpartum Period
Keywords: Performance; Servicewomen; Musculoskeletal; Well-Being

STUDY DESIGN:
Intervention Model Description: An independent group design with participants at one site receiving usual care/no formal intervention (acting as a control group [CON]) and participants at a second site receiving usual care and additionally completing an 18-week phased physical development (rehabilitation and training) programme between weeks 6 and 24 postpartum (acting as the intervention group [INT]).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Intervention (Experimental): 18-week physical development programme to train both rehabilitative and performance enhancement elements of physical preparation.
  Interventions: Other: Training intervention.
- Usual care control (No Intervention): Usual care acting as a control group.

INTERVENTIONS:
Other: Training intervention. — The investigators have designed a phased 18-week physical development programme to train both rehabilitative and performance enhancement elements of physical preparation. The rehabilitation element of the programme will specifically target pelvic floor function and core strength and stability (known collectively as Core Reconnection training) from weeks 6 to 24 postpartum, and the training element of the programme will contain resistance and high-intensity interval training (HIIT) from weeks 12 to 24 postpartum.
  Arms: Training Intervention

SUMMARY:
The purpose of this research is to investigate the effectiveness of a personalised physical training programme in returning servicewomen to fitness following childbirth. The idea behind the program is to target core and pelvic floor muscles, along with whole body strength and endurance to help servicewomen return to work safely and in a physically fit condition. The study will monitor the response to training using the following measures: urogynaecological measures (e.g., pelvic floor strength, prolapse, urinary incontinence), military specific fitness tests, musculoskeletal health (e.g., muscle and bone mass & function) and mental health and wellbeing.

DETAILED DESCRIPTION:
In an independent groups study design, the aim was to investigate the efficacy of a postpartum physical development programme on core reconnection (i.e., pelvic floor function, core strength/stability and urogynaecological measures), occupational physical performance, musculoskeletal health, and psychological health/wellbeing in servicewomen. Given that policy guidance is urgently needed regarding the safe return of servicewomen to functional occupational fitness, the aim of our proposed research is to inform the appropriate physical preparation of servicewomen in the postpartum period.

Participants at selected sites around the Royal Military Academy at Sandhurst will receive usual care/no formal intervention (acting as a control group [CON]) and participants at different sites around Army Headquarters will receive usual care and additionally complete an 18-week phased physical development (rehabilitation and training) programme between weeks 6 and 24 postpartum (acting as the intervention group [INT]). If recruitment numbers are low at the main sites (Aldershot and Tidworth) we will seek to recruit participants to INT from Bulford, Middle Wallop, Larkhill and Marlborough Lines for INT and to CON from Sandhurst, Odiham, Pirbright, Keogh, Minley, Deepcut as well as locations outside of the named INT sites. The geographical separation of sites was deemed to be important for maintaining differences between intervention and control group activity.

The investigators have designed a phased 18-week physical development programme to train both rehabilitative and performance enhancement elements of physical preparation. The rehabilitation element of the programme will specifically target pelvic floor function and core strength and stability (known collectively as Core Reconnection training) from weeks 6 to 24 postpartum, and the training element of the programme will contain resistance and high-intensity interval training (HIIT) from weeks 12 to 24 postpartum

The aim of this research is to investigate the effectiveness of a tailored rehabilitation and physical preparation programme for postpartum women on:

1. Occupational fitness performance;
2. Female health assessments (i.e., urinary incontinence, pelvic floor strength);
3. Musculoskeletal health;
4. Psychological health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

1. Serving, pregnant (third trimester) or 0 to 6 weeks postpartum UK MOD Servicewomen.
2. ≥ 18 years old.
3. Free from any condition or injury that may affect the individual's ability to perform exercise (health screen).
4. Passed fit to exercise by their GP at their routine 6-week postnatal check-up
5. Passed fit to participate by a specialist women's health physiotherapist using study specific assessment criteria.
6. Consent to be pregnancy tested before scans at 6 and 24 weeks postpartum.

Exclusion Criteria:

1. < 18 years old
2. Diagnosed with post-natal depression or another mental health condition requiring specialist psychiatric secondary care. Additionally, any participant who is found to have, or develops over the course of the trial, severe post-natal depression or suicidal tendencies, will be referred back to their GP.
3. Injured or suffering from another condition that can affect the individual's ability to perform exercise.
4. Not passed fit to exercise by their GP at their routine 6-week postnatal check [using standard fitness assessment criteria].
5. Not passed fit to participate following the women's clinical health assessment [using study specific assessment criteria].
6. Women who report that they could be pregnant and / or have a positive pregnancy test before measurements at 6 and 24 weeks postpartum will not be scanned using DXA or HR-pQCT. They will cease to take any further part in the trial and will be advised to visit their GP.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Physical Performance Change Between 12 and 24 Weeks Postpartum | Physical performance will be measured at weeks 12 and 24 postpartum.
  Physical performance will be measured at weeks 12 and 24 using elements of the Soldier Strength and Conditioning review , which the servicewomen need to complete as part of their return to service following maternity leave. These tests include a vertical jump, mid-thigh pull, seated medicine ball throw and a 2 km run to best effort.

SECONDARY OUTCOMES:
Pelvic Organ Prolapse- Quantification System Change in Scores Between 6, 12 and 24 Weeks Postpartum | : Pelvic Organ Prolapse- Quantification will be measured at weeks 6, 12 and 24 postpartum.
  Pelvic Organ Prolapse will be measured by the research associate women's health physiotherapist at weeks 6, 12 and 24. Vaginal examination will assess for prolapse using the Pelvic Organ Prolapse Quantification system staging pelvic support from 0-4, 0 being no prolapse demonstrated and 4 demonstrating full procidentia.
Pelvic Floor Strength Change in Scores Between 6,12 and 24 Weeks Postpartum | Pelvic floor distress inventory questionnaire will be measured at weeks 6, 12 and 24 postpartum.
  Pelvic floor strength will be measured by the research associate women's health physiotherapist at week 6, 12 and 24. Pelvic floor strength will be measured digitally using the modified oxford scale ranging from 0-5, 0 being no discernible contraction and 5 overcoming strong resistance. Over-activity and co-ordination of the pelvic floor muscle will be assessed by a simple yes/no answer following digital vaginal examination.
Musculoskeletal Physiotherapy Assessment Change Between 6,12 and 24 Weeks Postpartum | : Musculoskeletal physiotherapy assessment will be measured at weeks 6, 12 and 24 postpartum.
  Musculoskeletal physiotherapy measures will be assessed by the research associate women's health physiotherapist at weeks 6, 12 and 24. Posture, movement patterns, breathing will be objectively evaluated and commented on. The abdominal muscles (rectus diastasis) will be assessed by measuring the distance between the internal borders of the rectus abdominus muscle by placing the fingers vertically on the linea alba 4 cm above and below the umbilicus, during a curl up movement. Scoring is obtained through an approximation of centimetre width separation and the tone of the linea alba structure. The larger the score in centimetres the greater the separation of the rectus abdominus muscle.
Pelvic Floor Distress Inventory Questionnaire, Change in Scores Between 6, 12 and 24 Weeks Postpartum | Pelvic floor distress inventory questionnaire will be measured at weeks 6, 12 and 24 postpartum.
  The Pelvic Floor Distress Inventory will be completed at 6, 12 and 24 weeks by all participants. The Pelvic Floor Distress Inventory is scored ranging from 0-300, 0 being the least distress and 300 being the greatest distress.
International Consultation on Incontinence Questionnaire - Vaginal Symptoms, Change in Scores Between 6, 12 and 24 Weeks Postpartum | International consultation on incontinence questionnaire - vaginal symptoms will be measured at weeks 6, 12 and 24 postpartum.
  The International Consultation on Incontinence Questionnaire - Vaginal Symptoms will be completed at 6, 12 and 24 weeks by all participants. The International consultation on Incontinence Questionnaire - Vaginal Symptoms evaluates vaginal symptoms, associated sexual matters and impact on quality of life. Three scores are generated. Subscales range from 0-53 vaginal symptoms, 0-58 sexual matters and 0-10 overall impact on quality of life. 0 represents the least bothersome in each subscale. The subscales are not incorporated in an overall score.
World Health Organisation Quality of Life Questionnaire, Change in Scores Between 6, 12 and 24 Weeks Postpartum | The World Health Organisation Quality of Life Questionnaire will be measured at weeks 6, 12 and 24 postpartum.
  The World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF) will be given to participants in paper. The WHOQOL-BREF provides an overall quality of life/wellbeing score and allows calculation of a score for each of the four sub-scales (physical health, psychological, social relationships and environment). The four domain scores are scaled in a positive direction (higher score equal higher quality of life). The mean score of items within each domain is used to calculate the domain score.
Edinburgh Post Natal Depression Scale, Change in Scores Between 6, 12 and 24 Weeks Postpartum | The Edinburgh Post Natal Depression Scale will be measured at weeks 6, 12 and 24 postpartum.
  The Edinburgh Post Natal Depression Scale (EPDS) asks participants to answer questions by reflecting on the past 7 days. The questionnaire produces a total score of postnatal depression symptoms (range 0-30) with a score of 13 and above indicating likelihood of a depressive illness of varying severity
Body Composition Changes Between 6 and 24 Weeks Postpartum | Body composition will be measured at weeks 6 and 24 postpartum.
  Body composition (fat mass, fat-free mass and bone mineral density) will be measured at weeks 6 and 24 by a whole-body dual-energy x-ray absorptiometry (DXA) scan.
Bone Health Changes Between 6 and 24 Weeks Postpartum | Bone health will be measured at weeks 6 and 24 postpartum.
  Bone microarchitecture will be determined at weeks 6 and 24 by a HRpQCT scan; two scans of the tibia (distal 4% and 30% site) will be performed on the non-dominant leg to assess training-induced changes in bone microarchitecture and density.
Tendon Properties Changes Between 6, 12 and 24 Weeks Postpartum | Tendon properties will be measured at weeks 6, 12 and 24 postpartum.
  Tendon stiffness and young's modulus will be measured using ultrasonography with a linear array probe. Patella tendon length and elongation will be calculated as the distance from the apex of the patellar and the shadow created by a fixed marker. Patella tendon stiffness will be calculated by dividing knee extensor torque by the estimated patella tendon moment arm. Knee extensor torque will be calculated as the sum of the measured knee extension torque and the antagonistic torque, estimated through the root mean square of the biceps femoris muscle electromyography signal. Force-elongation data will be fitted with to a second order polynomial curve to determine patella tendon stiffness. Tendon CSA will be assessed along the full resting length of the tendon on the axial plane through ultrasonography. Young's modulus will then be calculated as tendon stiffness multiplied by the ratio of tendon length over tendon cross-sectional area.
Muscle Architecture Changes Between 6, 12 and 24 Weeks Postpartum | Muscle architecture will be measured at weeks 6, 12 and 24 postpartum.
  Fascicle length of the vastus lateralis will be assessed at weeks 6, 12 and 24 by the acquisition and analysis of images taken using B-mode ultrasonography (MyLab Omega, Esaote, UK), with a linear array probe. Images will be obtained with the participant lying at rest in a supine position. Images will be taken at 50% of the length of the vastus lateralis and at the midsagittal line of the muscle. The transducer will be aligned to the fascicle plane to allow optimal capture of the fascicles.
Muscle Protein and Collagen Turnover Changes Between 12 and 18 Weeks Postpartum | : Muscle protein and collagen turnover will be measured at weeks 12 and 18 postpartum.
  Muscle protein/collagen turnover will be measured from blood, saliva and skeletal muscle biopsy samples. Participants will provide a saliva sample before being given a drink of 'heavy' water (D2O); water that is enriched with a metabolic isotope tracer that can be used to evaluate the rate of protein and collagen turnover by determining the rate of tracer incorporation into muscle tissue. The muscle biopsy will be used to measure the incorporation of deuterated alanine into muscle tissue over time and enable the calculation of the fractional rate of muscle protein synthesis by mass spectrometry.
Muscle Mass Changes Between 6, 12, 18 and 24 Weeks Postpartum | Muscle mass will be measured at weeks 6, 12,18 and 24 postpartum.
  We intend to estimate whole-body muscle mass using D3-Creatine (D3-Cr), measured in urine at weeks 6, 12, 18 and 24 postpartum. Using a creatine-tracer measure of muscle mass, Urine D3-creatine and D3-creatinine and unlabelled creatine and creatinine will be measured by liquid chromatography/mass spectrometry, which will allow the calculation of total body creatine pool size and muscle mass.
Muscle Breakdown Changes Between 12 and 18 Weeks Postpartum | Muscle breakdown will be measured at weeks 12 and 18 postpartum
  We intend to estimate muscle breakdown using D3-3-methylhistidine (D3-3MH), measured in urine at weeks 12 and 18 postpartum. Isotopic enrichment of D3-3MH in urine will be measured by gas chromatography/mass spectrometry, which will allow the calculation of muscle protein breakdown.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Sale, PhD, Principal Investigator — Nottingham Trent University; Kirsty Elliott-Sale, PhD, Principal Investigator — Nottingham Trent University
Locations (11):
- United Kingdom (11):
  - Aldershot Centre for Health,, Aldershot, Hampshire,
  - Keogh Barracks, Aldershot, Hampshire
  - Station Medical Centre, Hook, Hampshire
  - Middle Wallop Medical Centre,, Stockbridge, Hampshire
  - MRS Royal Military Academy, Camberley, Surrey,
  - Minley Medical Centre, Blackwater, Surrey
  - The Princess Royal Barracks, Deepcut, Surrey
  - Elizabeth Barracks, Pirbright, Surrey
  - Larkhill Medical Centre, Salisbury, Wiltshire
  - Bulford Medical Centre, Salisbury, Wiltshire
  - Queen Elizabeth Memorial Health Centre, Tidworth, Wiltshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elliott-Sale KJ, Bostock EL, Jackson T, Wardle SL, O'Leary TJ, Greeves JP, Sale C. Investigating the Efficacy of an 18-Week Postpartum Rehabilitation and Physical Development Intervention on Occupational Physical Performance and Musculoskeletal Health in UK Servicewomen: Protocol for an Independent Group Study Design. JMIR Res Protoc. 2022 Jun 1;11(6):e32315. doi: 10.2196/32315. PMID 35648463